CLINICAL TRIAL: NCT05943795
Title: A Phase III Clinical Study of SI-B001 Combined With Docetaxel Second-line Therapy in Patients With Non-small Cell Lung Adenocarcinoma and Lung Squamous Cell Carcinoma Without Actionable Genomic Alterations Who Failed Only First-line Treatment With PD-1/PD-L1 Monoclonal Antibody Plus Platinum-Based Chemotherapy
Brief Title: A Clinical Study of SI-B001 Combined With Docetaxel in the Treatment of Non-small Cell Lung Adenocarcinoma and Lung Squamous Cell Carcinoma
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sichuan Baili Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SI-B001-301
Record Dates: First submitted 2023-04-04; First posted 2023-07-13 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Non-small Cell Lung Adenocarcinoma; Squamous Cell Carcinoma of Lung
MeSH Terms: interventions — Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Participants receive SI-B001 as intravenous infusion for the first cycle (3 weeks). Participants with clinical benefit could receive additional treatment for more cycles. The administration will be terminated because of disease progression or intolerable toxicity occurring or other reasons.
  Interventions: Drug: SI-B001
- Control group (Experimental): Participants receive Docetaxel as intravenous infusion for the first cycle (3 weeks). Participants with clinical benefit could receive additional treatment for more cycles. The administration will be terminated because of disease progression or intolerable toxicity occurring or other reasons.
  Interventions: Drug: Docetaxel

INTERVENTIONS:
Drug: SI-B001 — Administration by intravenous infusion
  Arms: Experimental group
Drug: Docetaxel — Administration by intravenous infusion
  Arms: Control group

SUMMARY:
Main objectives: To evaluate the benefit of SI-B001+ docetaxel on overall survival (OS) of bidotaxel. To evaluate the benefit of SI-B001+ Docetaxel over Docetaxel's progression-free survival (PFS) based assessment. Secondary objectives: To evaluate the investigator-evaluated progression-free survival (PFS) benefit of SI-B001+ Docetaxel against docetaxel; To evaluate the difference of objective response rate (ORR), disease control rate (DCR) and duration of response (DOR) between SI-B001+ docetaxel and bidocetaxel. To evaluate the type, frequency and severity of adverse events (TEAE) and drug-related adverse events (TRAE) during treatment with SI-B001+ docetaxel in comparison with docetaxel. The pharmacokinetic (PK) characteristics of SI-B001 will be evaluated. The immunogenicity of SI-B001 will be evaluated. Subject quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. Sign the informed consent form voluntarily and follow the protocol requirements;
2. Gender is not limited;
3. Age ≥18 years old and ≤80 years old;
4. Expected survival time ≥3 months;
5. Patients with histologically or cytologically confirmed locally advanced or metastatic non-small cell lung cancer;
6. Subjects had to consent to complete ctDNA testing during the screening period;
7. At least one measurable lesion meeting the RECIST v1.1 definition was required;
8. ECOG 0 or 1;
9. The toxicity of previous antineoplastic therapy has returned to ≤ grade 1 as defined by NCI-CTCAE v5.0;
10. No severe cardiac dysfunction, left ventricular ejection fraction ≥50%;
11. No blood transfusion is allowed within 14 days before the first use of the study drug, and the organ function level must meet the requirements on the premise that albumin and colony-stimulating factor are not allowed;
12. Coagulation function: international normalized ratio (INR) ≤1.5, and activated partial thromboplastin time (APTT) ≤1.5×ULN;
13. Proteinuria ≤2+ or < 1000mg/24h;
14. For premenopausal women with childbearing potential, a pregnancy test must be performed within 7 days before starting treatment, serum pregnancy must be negative, and the patient must not be lactating; All enrolled patients (male or female) were advised to use adequate barrier contraception throughout the treatment cycle and for 6 months after the end of treatment.

Exclusion Criteria:

1. Patients with previous docetaxel use;
2. Patients with non-small cell lung cancer (NSCLC) confirmed by histology or cytology except lung squamous cell carcinoma and lung adenocarcinoma;
3. The patients had received chemotherapy or biological therapy within 4 weeks or 5 half-lives before the first dose, and had received palliative radiotherapy or modern traditional Chinese medicine approved by NMPA for anti-tumor treatment within 2 weeks;
4. The history of severe cardiovascular and cerebrovascular diseases within six months before screening;
5. Prolonged QT interval, complete left bundle branch block, III degree atrioventricular block, frequent and uncontrollable arrhythmia;
6. Complicated with pulmonary diseases leading to severe impairment of lung function;
7. Active autoimmune and inflammatory diseases;
8. Other malignancies diagnosed within 5 years before the first dose;
9. Hypertension poorly controlled by two antihypertensive drugs (systolic blood pressure > 150 mmHg or diastolic blood pressure > 100 mmHg);
10. Patients with previous or current clinical manifestations or high risk factors such as ILD, drug-associated pneumonia, and radiation pneumonitis;
11. With untreated central nervous system metastases and/or carcinomatous meningitis/or spinal cord compression;
12. Patients with a history of allergy to the recombinant humanized or human-mouse chimeric antibody or to SI-B001 or any of the excipients of the chemotherapy drugs used in this trial;
13. Had a history of autologous or allogeneic stem cell transplantation or organ transplantation;
14. Human immunodeficiency virus antibody positive, active hepatitis B virus infection or hepatitis C virus infection;
15. Serious infection within 4 weeks before the first dose of study drug;
16. Pleural, pericardial, or abdominal effusion requiring drainage and/or associated with symptoms within 4 weeks before the first dose of study drug;
17. Received other investigational drugs or treatments within 4 weeks before the first dose;
18. A history of severe neurological or psychiatric illness;
19. Imaging examination showed that the tumor had invaded or wrapped the large thoracic vessels or pericardium or heart;
20. Serious unhealed wound, ulcer or fracture within 4 weeks before signing the informed consent;
21. Patients had hemoptysis or hemoptysis within 4 weeks before signing the informed consent, but those with blood in sputum were not excluded;
22. Had severe infusion reactions (CTCAE grade ≥3) to antibody therapy;
23. Subjects with clinically significant bleeding or obvious bleeding tendency within 4 weeks before signing the informed consent;
24. History of intestinal obstruction, inflammatory bowel disease, extensive bowel resection or chronic diarrhea;
25. Who are scheduled to receive the live vaccine or who receive it within 30 days before the first dose;
26. The investigator did not consider it appropriate to apply other criteria for participation in the trial.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 589 (Actual)
Dates: Start 2023-07-14 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) | Up to approximately 24 months
  Overall survival (OS) is defined as the time between the subject's randomization date and subject's death.
Progression-free survival (PFS) | Up to approximately 24 months
  Progression-free survival (PFS) as assessed by BIRC was defined as the time between the date subjects were randomized and the first observation of disease progression (based on BICR's image-based assessment) or death.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Up to approximately 24 months
  Objective response rate (ORR) is defined as the number of CR and PR in the treatment and control groups divided by the number of that group in the full analysis set (FAS).
Disease Control Rate (DCR) | Up to approximately 24 months
  Disease Control Rate (DCR) : Percentage of all randomized subjects who rated the best overall response (BOR) as complete response (CR), partial response (PR), and disease stabilization (SD) according to RECIST 1.1 criteria.
Duration of Response (DOR) | Up to approximately 24 months
  Duration of Response (DOR) : defined as the period from the date when tumor response is first recorded to the date when objective tumor progression is first recorded or the date of death.
Treatment Emergent Adverse Event (TEAE) | Up to approximately 24 months
  TEAE is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally emerging, or any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a pre-existing condition during the treatment of SI-B001. The type, frequency and severity of TEAE will be evaluated during the treatment of SI-B001.
Anti-drug antibody (ADA) | Up to approximately 24 months
  Characteristics of ADA will be evaluated.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang